CLINICAL TRIAL: NCT02171520
Title: Bioequivalence of Two Different Generations of Drug Product of 150 mg Dabigatran Etexilate Following Oral Administration in Healthy Male and Female Volunteers (Double-blind, Randomised, Single Dose, Replicate Design in a Two Treatments, Four Periods Crossover Phase I Study)
Brief Title: Bioequivalence of Two Different Generations of Drug Product of Dabigatran Etexilate Following Oral Administration in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.70
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- Dabigatran etexilate generation I (Experimental)
  Interventions: Drug: Dabigatran etexilate generation I
- Dabigatran etexilate generation II (Active Comparator)
  Interventions: Drug: Dabigatran etexilate generation II

INTERVENTIONS:
Drug: Dabigatran etexilate generation I
  Arms: Dabigatran etexilate generation I
Drug: Dabigatran etexilate generation II
  Arms: Dabigatran etexilate generation II

SUMMARY:
The objective was to demonstrate the bioequivalence of capsules made from 2 different drug product batches. The reference batch was representative of the current commercial drug product and of the pivotal Phase III batches. The test batch was the drug product batch intended for future commercial use.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, clinical laboratory tests
2. Age ≥60 and ≤85 years
3. Body mass index (BMI) ≥18.5 and BMI ≤30.0 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Clinically relevant surgery of gastrointestinal tract
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. Any relevant bleeding history
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within four weeks prior to administration or during the trial
11. Alcohol abuse (more than 60 g/day for men and more than 40 g/day for woman)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance (especially hemoglobin and activated partial thromboplastin time) or positive drug or virus screening
16. Planned surgeries within four weeks following the end-of study examination
17. Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
18. Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
19. Subject is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study
20. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, coumarin etc. within 10 days prior to administration
21. Vulnerable subjects (e.g. persons kept in detention)
22. Male subjects who do not agree to minimise the risk of female partners becoming pregnant from the first dosing day until the completion of the post study medical examination. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two months)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 extrapolated to infinity) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
Cmax (maximum measured concentration of total dabigatran in plasma) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 extrapolated to infinity) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
Cmax (maximum measured concentration of free dabigatran in plasma) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
AUCt1-t2 (area under the concentration time curve of the analyte in plasma over the time interval t1 to t2 with t1 = 0 and t2 = 24, 48, 72 hours) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
λz (terminal rate constant in plasma) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
t1/2 (terminal half-life of the analyte in plasma) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | before drug administration and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours following drug administration